CLINICAL TRIAL: NCT04626830
Title: The Effect of a Mobile Application on Treatment Adherence and Symptom Management in Patients Using Oral Anticancer Agents: A Randomized Controlled Trial
Brief Title: Mobile Application to Assist Adherence to Oral Anticancer Agents and Symptom Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Koç University (Other); Gazi University (Other)
Responsible Party: Principal Investigator, Akile Karaaslan Eşer, Assistant professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Project No: 2018.1.18.
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Adherence to Medication Regime; Symptom Management
Keywords: Cancer; Mobile applications; Oral anticancer agents; Oral Chemotherapy; Medication adherence; Nursing
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Intervention (Experimental): Participants in the intervention group will receive 6 months the mobile application (OKTED) for improving symptoms and adherence to oral anticancer agents. The mobile application will consist of three modules. The first module will include OAA-specific information, a calendar in which start/end dates can be record, and a medication reminder. The second module will include information about common and urgent symptoms and recommendations for the management of these symptoms. The last module will comprise a question and answer section.
  Interventions: Other: Mobile Application Intervention
- Standard Care (No Intervention): Participants in the control group will receive standard oncology care only.

INTERVENTIONS:
Other: Mobile Application Intervention — Participants appointed to the intervention group will receive the mobile application intervention for six months after enrollment. The mobile app (OKTED) intervention will consist of completing responding to weekly assessments regarding symptoms, side effects, and medication adherence, as well as receiving personalized feedback about responses.
  Arms: Mobile Application Intervention

SUMMARY:
The use of oral anticancer agents (OAAs) in cancer treatment has increased especially in the last two decades. The use of mobile health technologies in the management of OAA can be beneficial in terms of treatment adherence and symptom management.The aim of this study is to explore how a Smartphone mobile application can help improve the cancer treatment process in people who are used oral anticancer agents. This study will be done a randomized-controlled trial to test the intervention.

DETAILED DESCRIPTION:
Background: The use of mobile health technologies in the management of OAA can be beneficial in terms of treatment adherence and symptom management.

Objective/Hipothesis: The purpose of this study is to explore the effectiveness of a mobile application on treatment adherence and symptom management in patients using OAA. The following hypotheses (H) will teste in this study:

H0a: A mobile application developed for patients using OAA has not increased treatment adherence.

H1a: A mobile application developed for patients using OAA has increased treatment adherence.

H0b: A mobile application developed for patients using OAA has not decreased the frequency and severity of symptoms.

H1b: A mobile application developed for patients using OAA has decreased the frequency and severity of symptoms.

Study Design: The investigators will recruit and randomly assign 100 patients from the two cancer care sites who have recently been prescribed oral anticancer agents to receive either the mobile app intervention or standard care. Participants will be stratified by age and anticancer treatment ( i.e. simple and complex) regimen. Patients will be follow 6 months. Medication adherence, symptom severity will serve as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Using OAAs for cancer treatment and taking at least one cure
* Taking OAAs for at least six months
* Knowing the diagnosis
* Communicating verbally
* Scoring less than three on the Eastern Cooperative Oncology Group (ECOG) scale
* Having a smartphone with IOS or Android software
* Actively using the smartphone
* Consenting to download the mobile application on one's mobile phone
* Volunteering to participate in the research.

Exclusion Criteria:

* Participation in a similar study aimed at increasing treatment adherence
* Having physical, cognitive, or memory-related problems that significantly impair one's daily activities
* Having a smartphone with Windows or Blackberry software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to Oral Anticancer Agents | baseline, 1 month, 3 months, 6 months
  The patients' adherence levels will be assess using the Oral Chemotherapy Adherence Scale (OCAS). The OCAS was developed by Bagcivan and Akbayrak (2015), and its Cronbach α coefficient was found to be 0.738. The scale (19 items, 5-point Likert-type) is a valid and reliable scale for adult patients who use OAAs. A total score of 84 and above is interpreted as "good adherence;" a total score of 83 and below is interpreted as "poor adherence".
Change in Symptoms and Side Effects | baseline, 1 month, 3 months, 6 months
  The Memorial Symptom Assessment Scale (MSAS) is a multidimensional tool developed to evaluate the prevalence, characteristics, and distress levels of common cancer-related symptoms over seven days (Cronbach α=0.84). The MSAS is a reliable and valid instrument in the Turkish population. The scale has 32 items and three sub-dimensions: The Global Distress Index, The Physical Symptom Distress Scores, and The Psychologic Symptom Distress Scores. The total MSAS score is the average of the symptom scores of all 32 items. Twenty-four symptoms are evaluated in terms of severity, frequency and distress, and eight symptoms are evaluated in terms of severity and distress. If a symptom was experienced, the patient describes its severity on a 4-point categorical scale; its frequency, if appropriate, on a 4-point categorical scale; and its associated distress on a 5-point categorical scale. Each symptom score is the average of the dimensions (frequency, severity, distress dimensions).

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karaaslan-Eser A, Ayaz-Alkaya S. The effect of a mobile application on treatment adherence and symptom management in patients using oral anticancer agents: A randomized controlled trial. Eur J Oncol Nurs. 2021 Jun;52:101969. doi: 10.1016/j.ejon.2021.101969. Epub 2021 May 4. PMID 33991868